CLINICAL TRIAL: NCT03898817
Title: Pathology of Helicases and Premature Aging: Study by Derivation of hiPS
Acronym: HeliPS
Status: Terminated | Type: Observational
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9360
Record Dates: First submitted 2016-09-07; First posted 2019-04-02 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Age Problem
Keywords: helicase; induced pluripotent stem cells

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Taking of cutaneous cells by biopsy: Taking of cutaneous cells by biopsy and a sample of blood
  Interventions: Other: taking of cutaneous cells

INTERVENTIONS:
Other: taking of cutaneous cells — Taking of cutaneous cells by biopsy Sample of blood

SUMMARY:
Topic of this work is the involvement of replicative helicases in human premature ageing syndrome. Replicative helicases are ubiquitous and essential during numerous reactions of the DNA metabolism.

The family of replicative helicases (RecQL) is involved in the replication/repair of the DNA and in the telomere maintenance. There are 5 enzymes in human and 3 of them are involved in clinically recognizable syndromes: WRN for the Werner syndrome, BLM for the Bloom syndrome and RECQL4 for the Rothmund Thomson syndrome. All are responsive of a high cancer risk due to genomic instability. Molecular and cellular mechanisms involved in these diseases of ageing are unknown. Moreover, for all of them, there is not therapeutic or preventive solution.

DETAILED DESCRIPTION:
For understanding the involved mechanisms we would like to model the 3 diseases with hiPS (human induced Pluripotent Stem cells) from somatic cells of patients. The patient recruitment was organized by the Montpellier and Nîmes public hospitals.

The project is to generate a hiPS cell line for the 3 syndromes from fibroblasts and/or blood samples. Then, we could induce differentiation of hiPS to a target cell line of the diseases. Finally we could study the disease development following the genomic instability (karyotype, array-CGH) and the cellular ageing (senescence-associated heterochromatin foci, telomere length).

For each mutated enzyme, we will perform a transcriptional profiling (splice, mRNA quantification) and protein studies (western blot). All results will be compared to wild type cells.

ELIGIBILITY:
Inclusion Criteria:

* Patinet with one of the 3 helicase-associated precoce aging desease

Exclusion Criteria:

* Minor and /or mentally incapable patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with pathology of helicases and premature aging
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2017-09-09 (Actual)

PRIMARY OUTCOMES:
Genomic instability : analysis | 1 year
  Molecular analysis of hiPS cell derived from pathological tissue (karyotype, array-CGH)
Genomic instability : size of telomers | 1 year
  size of the telomers which will be quantified under microscope after fluorescent marking in situ of telomeric sequences (Q-FISH technique)
Genomic instability : Duplication of centrosomes | 1 year
  duplication of centrosomes which is often associated with chromosomal segregation errors and genomic instability. This analysis will be done by immunolabelling using antibodies specific to the 2 main components of centrosomes, pericentrin and -tubulin.

SECONDARY OUTCOMES:
cellular ageing : molecular analysis of hiPS cell derived from pathological tissue | 2 years
  Analysis of senescence-associated heterochromatin foci, telomere length (Q-FISH)
cellular ageing : IPS line with the criteria defined for morphological characterization | 2 years
  expression of specific surface markers (specifics markers : TRA-1-60, SSEA-4), ability to re-differentiate in the 3 embryonic layers (specifics markers : SMA, MAP2, FOXA2)
cellular ageing : molecular characterization | 2 years
  lengthening of telomeric sequence size (Q-FISH), re-expression of pluripotency genes (QRTPCR), transcriptional profile of iPS cell lines.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GATINOIS, harmD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No